CLINICAL TRIAL: NCT02505620
Title: Neurocognitive Function After Surgical and Conservative Therapy in OSAS Patients: a Randomized Control Trial
Brief Title: Neurocognitive Function After Therapy of OSAS
Acronym: 203_14_B
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2015-06-09; First posted 2015-07-22 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Neurocognitive Function; OSAS
Keywords: Neurocognitive function; OSAS
MeSH Terms: interventions — Continuous Positive Airway Pressure; Masks; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical: Surgical correction of OSAS disease
  Interventions: Procedure: Surgical Treatment with multilevel operation
- Conservative: Conservative treatment of OSAS disease
  Interventions: Procedure: Treatment of OSAS with CPAP mask

INTERVENTIONS:
Procedure: Treatment of OSAS with CPAP mask — Interventional treatment addresses the treatment with a CPAP (continuous positive airway pressure) mask in oder to open patients upper airway obstructive permanently while sleep.
  Other Names: CPAP (continuous positive airway pressure) mask
  Groups: Conservative
Procedure: Surgical Treatment with multilevel operation — Surgical treatment addresses a surgical multilevel anti-obstructive operation in order to eliminate upper airway obstruction permanently.
  Other Names: Surgical multilevel anti-obstructive operation
  Groups: Surgical

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is characterized by repeated episodes of airway obstruction while sleeping. Upper airway obstruction while sleeping leads to a dramatic decrease in oxygen saturation and to hypoxemia finally, in which consequence the patient rapidly awake. Clinical signs are sleepiness and functional cognitive deficits. The Gold standard therapy is "continuous positive airway pressure" ventilation during sleep. However, the success depends strongly to the patient´s compliance. Surgical treatment is an alternative option, which could be considered if clinical success failed. A comparison of the cognitive function of both therapies is not yet analyzed. The study addresses the question which of this treatment options is favorable regarding cognitive function and outcome.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome (OSAS) is characterized by repeated episodes of airway obstruction while sleeping. The "Apnea-hypopnea index" (AHI) defined as events per hour, gives information about the severity of the disease. The American Academy of Sleep Medicine Task Force" defined that more than 5 episodes per hour is strongly suspect for an OSAS disease. Upper airway obstruction while sleeping leads to a dramatic decrease in oxygen saturation and to hypoxemia finally, in which consequence the patient rapidly awake. The prevalence rise with age and about 20% of the population is suspect to a sleep disorder. However about 1-5% of male and about 0,5-2% of female aged adults are affected. Main reason is obesity. Clinical signs are sleepiness and functional cognitive deficits. The Gold standard therapy is "continuous positive airway pressure" ventilation during sleep. However, the success depends strongly to the patient´s compliance. Surgical treatment is an alternative option, which could be considered if clinical success failed. It is notable that the long-term mortality is comparable in both medical treatment options. However, a comparison of the cognitive function of both therapies is not yet analyzed. The study addresses the question which of this treatment options is favorable regarding cognitive function and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 30 to 70 years of age both gender.

Exclusion Criteria:

* Patients under 30 years of age or older than 70 years of age.
* Preexisting neurological, neuropsychological deficits or diseases, e.g. cerebral insult or epilepsy.
* Preexisting neurological, neuropsychological medication.
* Preexisting neuromuscular diseases.
* Alcohol - and drug abuse.
* Postoperative complications, pain and time shifts within the test protocol.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruted at the University Hospital Erlangen prior surgery or conventional treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function | 4 months
  Using different tests addressing a various quality of neurocognitive function (attention, memory, perceptual and processing speed, alertness and executive function) participants score test appropriate values. Comparing test values separately allows to distinguish between prior - and post - operative and prior and post - interventional status. Moreover it allows to discriminate achieved test results between both groups and calculate statistical differences. Favorable test results lead to a potential better neurocognitive function outcome and enable to assess neurocognitive function in the light of operation or interventional consequence.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Dept. Anaesthesiology, Erlangen, Germany